CLINICAL TRIAL: NCT03910361
Title: A Multicenter, Double-blind, Active-controlled, Randomized, Parallel, Phase IV Clinical Trial to Evaluate the Efficacy and Safety of Evogliptin in Patients With Type 2 Diabetes and Non-alcoholic Fatty Liver Diseases
Brief Title: Efficacy and Safety of Evoglitin in Patients With Type 2 Diabetes and Non-alcoholic Fatty Liver Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA1229_NAFLD_IV
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Type2 Diabetes; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evogliptin (Experimental): evogliptin 5mg
  Interventions: Drug: Evogliptin
- Pioglitazone (Active Comparator): pioglitazone 15mg
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Evogliptin — evogliptin 5mg tablet qd + placebo tablet matching to pioglitazone 15mg qd
  Other Names: Suganon
  Arms: Evogliptin
Drug: Pioglitazone — pioglitazone 15mg tablet qd + placebo tablet matching to evogliptin 5mg qd
  Other Names: Gluconon
  Arms: Pioglitazone

SUMMARY:
A multicenter, double-blind, active-controlled, randomized, parallel, phase IV clinical trial to evaluate the efficacy and safety of evogliptin in patients with type 2 diabetes and non-alcoholic fatty liver diseases

DETAILED DESCRIPTION:
1. Evogliptin 5mg Group: Administration with Evogliptin 5mg and Placebo for 24weeks
2. Pioglitazone 15mg Group: Administration with Pioglitazone 15mg and Placebo for 24weeks

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus
* Subjects who have not been taking any oral hypoglycemic agent within 8 weeks from screening or who have been taking metformin monotherapy at the same dose for more than 8 weeks before screening
* Subjects with 6.5%≤HbA1c≤9.0% at screening
* Subjects with 20kg/m2≤BMI≤40kg/m2 at screening

Exclusion Criteria:

* Type I diabetes mellitus, secondary diabetes mellitus or gestational diabetes mellitus
* AST > upper normal range*3
* Galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Subjects who experienced hypersensitivity reaction against DPP-4 inhibitors, thiazolidinediones
* Pregnant women

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Changes from baseline intrahepatic fat (%) | 24 weeks
  Changes from baseline intrahepatic fat (%) after treatment with evogliptin or pioglitazone

CONTACTS AND LOCATIONS:
Overall Officials: Byung Wan Lee, Principal Investigator — Severance Hospital
Locations (7):
- South Korea (7):
  - Samsung Medical Center, Changwon
  - Soonchunhyang University Hospital, Cheonan
  - Keimyung Dongsan University Medical Center, Daegu
  - Hanyang University Guri Hospital, Guri-si
  - Catholic University of Seoul ST.Mary's Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul